CLINICAL TRIAL: NCT06093009
Title: National Cheng Kung University Hospital
Brief Title: The Significance of Postoperative Muscle Wasting in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER-110-420
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreatectomy

SUMMARY:
To assess the impact of preoperative sarcopenia and postoperative skeletal muscle wasting on the outcomes of patients with resectable pancreatic cancer who underwent pancreatectomy.

DETAILED DESCRIPTION:
Previous studies have revealed that sarcopenia, defined as generalized loss of skeletal muscle mass, is a poor prognostic factor following surgery. However, research focusing on postoperative muscle wasting and its influence on the prognosis of resectable pancreatic cancer (PC) is limited. Investigators retrospectively reviewed 208 patients who underwent pancreatectomy for PC at the National Cheng Kung University Hospital (NCKUH) between June 2002 and April 2020. Clinical information regarding patient characteristics, pathological parameters, and biochemical features was collected from all patients using electronic medical records (EMRs) under an IRB-approved protocol (B-ER-110-420) at NCKUH. Preoperative psoas major area and the degree of muscle reduction at 3 months postoperatively were calculated using computed tomography to define sarcopenia and drastic muscle wasting. Patients were assigned to two groups based on sarcopenia or drastic muscle wasting, and compared for postoperative morbidity, disease free survival (DFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pancreatic cancer
* Must be able to undergo pancreatectomy
* Must be able to undergo pre- and post-operative abdominal computed tomography scan

Exclusion Criteria:

* Unresectable pancreatic cancer

Ages: 20 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 20 Years and older (Adult, Older Adult ).
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2002-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Overall survival was measured as the period between the date of resection and the date of the last follow-up or death.
Disease-free survival | 10 years
  Disease-free survival was defined as the duration from resection to cancer relapse (local, peritoneal recurrence, or distal metastasis).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to privacy issues.